CLINICAL TRIAL: NCT01471288
Title: Evaluation of the Effect of Carum Carvi on Levels of Plasma Thyroid Hormones and TSH Level in Patients on Thyroid Hormone Therapy and Normal Controls.
Brief Title: Effect of Carum Carvi on Thyroid Hormones and TSH Level
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Collaborators: Pharmaceutical Research Center (Unknown)
Responsible Party: Seyed Rasoul Zakavi, Nuclear Medicine Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 88498
Record Dates: First submitted 2011-07-21; First posted 2011-11-15 (Estimated); Last update posted 2011-11-15 (Estimated); Status verified 2011-10

CONDITIONS: Thyroid Cancer Patients
Keywords: well differentiated thyroid cancer; Carum Carvi; Normal controls

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group3 (Active Comparator): Normal controls
  Interventions: Drug: Carum Cravi
- Group4 (Placebo Comparator): Normal controls
  Interventions: Drug: Placebo
- Group 1 (Active Comparator): Hypothyroid patients taking levothyroxin.
  Interventions: Drug: Carum Cravi
- Group2 (Placebo Comparator): Hypothyroid patients taking levothyroxin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carum Cravi — 40mg/kg of body weight
  Arms: Group 1; Group3
Drug: Placebo — Placebo
  Arms: Group2; Group4

SUMMARY:
Carum Carvi has been frequently used in traditional medicine for a variety of disease ranging from dyspepsia to Alzheimer's disease.We observed high TSH levels in few patients with thyroid cancer who receiving Carum Carvi despite being on suppressive dose of levothyroxin. TSH level returned to normal after discontinuation of the Carum carvi. This observation led to a pilot study for evaluation of the effect of carum carvi on thyroid function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Hypothyroid patients under treatment with levothyroxin
* Normal euthyroid patients with no goiter

Exclusion Criteria:

* Pregnancy or lactation
* Severe lung or gasterointestinal disease
* Heart failure or renal failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Change of Thyroid and thyrotropin values from baseline at 2 and 6 weeks | 0-2-6 Weeks
  TSH, Free T4, Free T3, T4RIA and T3RIA

SECONDARY OUTCOMES:
Change of hypothyroidism index from baseline at 2 and 6 weeks | 0,2 and 6 weeks
  Hypothyroidism Index

CONTACTS AND LOCATIONS:
Overall Officials: Seyed Rasoul Zakavi, MD. IBNM, Principal Investigator — Nuclear Medicine Research Center; Mohammad Ramezani, Ph.D., Pharm.D, Principal Investigator — Pharmaceutical Research Center
Locations (1):
- Nuclear Medicine Department, Ghaem Hospital, Mashhad, Iran